CLINICAL TRIAL: NCT04302831
Title: Restoring Central Motor Control to Improve Community Mobility of Older Adults
Brief Title: Restoring Central Motor Control Extension
Acronym: PRIMA-NIRS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 safety restrictions
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Andrea Rosso, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY19110142; R01AG057671-01A1 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Gait, Unsteady
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): The standard arm consists of strength, endurance and flexibility exercises 2 times per week for 12 weeks. Will also receive a physical activity behavioral intervention.
  Interventions: Behavioral: Strength training; Behavioral: Endurance training; Behavioral: Flexibility training; Behavioral: Physical activity behavioral intervention
- Standard-plus (Experimental): The standard-plus arm consists of strength, endurance and flexibility exercises plus task specific timing and coordination exercises to improve gait 2 times per week for 12 weeks. Will also receive a physical activity behavioral intervention.
  Interventions: Behavioral: Strength training; Behavioral: Endurance training; Behavioral: Flexibility training; Behavioral: Physical activity behavioral intervention; Behavioral: Task Specific timing and coordination training

INTERVENTIONS:
Behavioral: Strength training — weight lifting to increase muscle strength
Behavioral: Endurance training — treadmill walking to increase endurance
Behavioral: Flexibility training — stretches to improve flexibility
Behavioral: Physical activity behavioral intervention — Intervention to encourage participants to be more physically active
Behavioral: Task Specific timing and coordination training — stepping and walking patterns to improve timing and coordination of gait
  Arms: Standard-plus

SUMMARY:
Motor skill training therapy aims to improve the brain's control of walking and can improve clinic-based measures of walking in older adults. However, it is unknown whether the benefits of motor skill training extend to real world mobility measures. The investigators will test the effects of motor skill training on measures of community mobility of older adults and assess the mechanisms through improved motor control at the level of the brain. These results will inform intervention approaches to maintain community mobility of older adults and prevent disability and institutionalization.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* Ambulatory without an assistive device or the assistance of another person
* Usual 4 meter gait speed > 0.60 m/s and < 1.2 m/s
* Physician clearance to participate in a moderate intensity exercise program
* Not meeting physical activity recommendations defined as reporting less than 150 minutes of moderate intensity activity per week in the past month.

Exclusion Criteria:

* persistent lower extremity pain that is present on most days of the week
* back pain that is present on most days of the weeks and interferes with walking and - activities of daily living or back pain that increases with walking
* refuse to walk on a treadmill
* plans to move out of the area in the next 5 years
* dyspnea at rest or during activities of daily living or use supplemental oxygen (CHF, COPD)
* any acute illness or medical condition that is not stable according to the approving physician
* resting systolic blood pressure ≥ 200 mm Hg or diastolic blood pressure ≥ 100 mm Hg or resting heart rate > 100 or < 40 beats per minute
* diagnosed dementia or cognitive impairment defined as modified Mini-Mental State (3MS) examination <79
* hospitalized in the past 6 months for acute illness or surgery, other than minor surgical procedures
* severe visual impairment f- ixed or fused lower extremity joints such as hip, knee or ankle
* lower extremity strength <3/5 on manual muscle testing
* lower extremity amputation
* progressive movement disorder such as Multiple Sclerosis, Amyotrophic Lateral Sclerosis or Parkinson's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in oxygenated hemoglobin at the prefrontal cortex from standing to walking | change from baseline to 12 weeks
  Physiologic measure indicative of usage of the prefrontal cortex during a task recorded by optical imaging (near infrared spectroscopy).
Change in oxygenated hemoglobin at the prefrontal cortex from standing to walking | change from baseline to 36 weeks
  Physiologic measure indicative of usage of the prefrontal cortex during a task recorded by optical imaging (near infrared spectroscopy).

SECONDARY OUTCOMES:
Gait speed | 12, 24, and 36 weeks
  Walking speed (m/s) during usual pace
Gait speed | 12, 24, and 36 weeks
  Walking speed (m/s) with a cognitive challenge.
Gait speed | 12, 24, and 36 weeks
  Walking speed (m/s) on an uneven surface.
Gait variability | 12, 24, and 36 weeks
  Fluctuations in gait characteristics from step to step during usual pace. Physiologic measure of temporal gait characteristics (standard deviation).
Gait variability | 12, 24, and 36 weeks
  Fluctuations in gait characteristics from step to step while walking with a cognitive challenge. Physiologic measure of temporal gait characteristics (standard deviation).
Gait variability | 12, 24, and 36 weeks
  Fluctuations in gait characteristics from step to step while walking on an uneven surface. Physiologic measure of temporal gait characteristics (standard deviation).

OTHER OUTCOMES:
Activity Space | 12, 24, and 36 weeks
  Extent of travel beyond the home collected by GPS device based on a standard deviation ellipse of spatial measurement points.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Rosso, PhD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No